CLINICAL TRIAL: NCT00758433
Title: Randomized, Double-Blind, Placebo-Controlled Evaluation of the Tolerability of Two Civamide (Zucapsaicin) Patch Strengths Compared to Placebo Patch in Healthy Volunteers
Brief Title: Civamide Patch Safety, Tolerability and PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Study Director, Winston Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: WL-1001-04-01
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers
Keywords: Adverse Events; Erythema Rating; Pharmacokinetics; Civamide; Phase 1; Pain; Patch
MeSH Terms: conditions — Pain | interventions — zucapsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Civamide patch 0.0075%
  Interventions: Drug: Zucapsaicin
- 2 (Active Comparator): Civamide patch 0.0150%
  Interventions: Drug: Zucapsaicin
- 3 (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Zucapsaicin — Civamide patch 0.0075% q.d. 24 hours for 7 days
  Other Names: Civamide
  Arms: 1
Drug: Zucapsaicin — Civamide patch 0.0150% q.d. 24 hours for 7 days
  Other Names: Civamide
  Arms: 2
Drug: Placebo patch — Placebo patch q.d. 24 hours for 7 days
  Other Names: placebo
  Arms: 3

SUMMARY:
To evaluate the tolerability of two different strengths of a Civamide Patch (0.0075% and 0.0150%) compared to the placebo patch and each other in healthy adult volunteers. To assess the pharmacokinetics of civamide and to determine if there is systemic absorption of the drug from civamide patch in a subset of study subjects.

DETAILED DESCRIPTION:
This is a double-blind, randomized study of the tolerability of two different strengths of a Civamide Patch compared to placebo patch. The study consists of a Screening Period (Days -21 to Day 1), a one week Treatment Period (Days 1-8) and a follow-up telephone call to subjects on Day 10.

Pharmacokinetics will be assessed relative to dosing on Day 1, Day 2, and Day 8 in a subset of subjects. Subjects will also rate stinging and burning sensation at the application site during the Treatment Period.

Twenty-four (24) hours after the last patch application, subjects will return to the study site on Day 8. The treatment area will be evaluated by the Study Physician. Subjects will complete a Subject's Global Rating of Stinging and Burning Sensation and a Subject's Global Rating of Tolerability.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Subject voluntarily agrees to participate in this study and signs an IRB- approved informed consent prior to performing any of the screening procedures.
2. Subject is healthy, determined by pre-study medical evaluation medical history, physical examination of the treatment area, and vital signs).
3. Males or females between 18 to 60 years of age, inclusive.
4. Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, or intrauterine device) from Screening to Day 10 follow-up or females of nonchildbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year).
5. Subject has a blood pressure reading lower than or equal to 144/92 mmHg.
6. Subject has an oral temperature reading lower than 99.6F.
7. Subjects must have an area of the skin on the abdomen that is without active skin disease, infection, severe erythema, or other compromise in the integrity of the skin at or near the intended treatment area.
8. The subject has no visual or motor impairments that will make it difficult to complete the VAS scales or apply the patch.
9. Non-smoker as determined by history over the past year.
10. Subject has a body mass index (BMI) between 18.5 and 30.5 kg/m2, in pk subset only.
11. Subject is willing and able to cooperate to the extent required by the protocol.

Exclusion Criteria:

1. Subject has known allergy or hypersensitivity to

   * a) Civamide, capsicum, or capsaicin-containing products,
   * b) any other ingredient of the patch or
   * c) adhesives.
2. Presence of any cutaneous abnormality or condition that may adversely impact the application of the test patches.
3. History of frequent headache or other painful conditions within the past 30 days that has required or is expected to require the chronic use of prescription or over the counter pain relief medications, such as non- steroidal anti-inflammatory agents, including COX-2 inhibitors, systemic opiates or derivatives, or acetaminophen, prior to Day 1 or within 48 hours prior to Day 1.
4. Use of alcohol or alcohol-containing foods, medications or beverages within 24 hours prior to Day 1 until after the completion of the Study on Day 10.
5. Topical use of any moisturizer or medicated products on or near the treatment area within 48 hours of Day 1 until after the completion of the Study on Day 10.
6. Topical use of any capsaicin-containing product for 60 days prior to Day 1 until completion of the Study on Day 10.
7. Subject has a history of alcohol and/or drug abuse within two years of study entry.
8. Female subjects who are breastfeeding.
9. Unwilling to maintain usual consumption of caffeine containing beverages within 24 hours prior to Day -1 until completion of Day 8.
10. Subject is unwilling to abstain from vigorous exercise for 48 hours prior to Day 1 until completion of the Study on Day 10.
11. Subject is unwilling to abstain from swimming, baths and prolonged with direct stream of water when showering from Day 1 until Day 8
12. Use of an investigational drug within 30 days prior to Day 1.
13. Donation of blood (> 250 ml) or blood products within 2 months (56 days) prior to Day 1.
14. Ingestion of any capsaicin-containing foods for 24 hours before Day 1 and during the study.
15. If for any other reason the subject is not deemed to be healthy by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Subject's Rating of Stinging and Burning Sensation | 7 Days

SECONDARY OUTCOMES:
Pharmacokinetics | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, M.D., Study Director — Winston Laboratories
Locations (1):
- International Research Services, Inc., Port Chester, New York, United States